CLINICAL TRIAL: NCT04855773
Title: Comparing Mobile Health Strategies to Improve Pre-exposure Prophylaxis Use (PrEP) for HIV Prevention
Acronym: PCORI PrEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of California, San Francisco (Other); University of Miami (Other); Whitman-Walker Health (Unknown); San Francisco AIDS Foundation (Other); WelTel (Unknown); San Francisco Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Albert Liu, Clinical Research Director, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-32976
Record Dates: First submitted 2021-04-01; First posted 2021-04-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Pre-exposure Prophylaxis (PrEP); HIV Prevention; Mobile health (mHealth); Medication adherence
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEPmate (Experimental): Participants randomized to this study arm will receive the PrEPmate mHealth intervention (bi-directional text messaging with PrEP navigators/clinic staff) to support PrEP adherence and continuation.
  Interventions: Other: PrEPmate
- Dot Diary mobile application (Experimental): Participants randomized to this study arm will download and use the Dot Diary mobile application on a personal device, to support PrEP adherence and continuation.
  Interventions: Device: Dot Diary

INTERVENTIONS:
Other: PrEPmate — PrEPmate is a multi-component mHealth intervention grounded in the information, motivation, behavioral skills (IMB) theory of behavior change and developed through user-centered design. PrEPmate promotes personalized communication between patients and providers through interactive weekly "check-in" messages asking participants how PrEP is going, allowing navigators to identify patients needing more help in taking PrEP, and customized daily pill-taking reminder messages. Trained PrEP navigators reach out to participants who indicate they need assistance via text or phone call and provide tailored support. Additionally, the platform supports 2-way communication between patients and PrEP navigators, including reminders for upcoming clinic visits. Participants are provided links to key information about PrEP (PrEP Basics), and video testimonials of peers taking PrEP. Messages are available in English and Spanish. PrEPmate is aimed at both patients and PrEP navigators.
  Arms: PrEPmate
Device: Dot Diary — Dot Diary is a mobile phone app that integrates an electronic pill-taking and sex diary and delivers real-time feedback on PrEP protection. Using the self-management model to increase self-efficacy and patient empowerment, participants log daily PrEP pill-taking and sexual behaviors in the app, which then provides real-time feedback on the level of protection achieved from PrEP (high, medium, low), and customized instructions on doses of PrEP needed to achieve or maintain high protection. Participants can also view a weekly and monthly calendar, including visualizations of the proportion of sex acts covered by PrEP. Finally, the Dot Diary app incorporates gamification components, including an ability to earn sex-positive badges, to increase engagement. Dot Diary is aimed only at patients.
  Arms: Dot Diary mobile application

SUMMARY:
The purpose of this study is to compare the effectiveness of two mobile health technologies (text messaging or a mobile app) designed to help people take HIV pre-exposure prophylaxis (PrEP) as directed by the clinic. PrEP is the use of a daily anti-HIV medications by HIV-negative people to help prevent HIV infection.

DETAILED DESCRIPTION:
This is a clinic-based, multi-site, randomized, two-arm study to compare the effectiveness of two mobile technologies designed to support PrEP adherence and continuation in cisgender and transgender men who have sex with men (MSM) and transgender women (TGW). All study participants will receive PrEP per standard of care at each of the study sites.

Participants randomized to PrEPmate will receive an interactive bidirectional text-messaging intervention that supports PrEP use through personalized communication between patients and providers. Key components include (1) weekly short message service (SMS) check-ins and a bidirectional SMS messaging platform; (2) customized daily SMS pill-taking reminders; (3) link to online PrEP Basics and videos and testimonials.

Participants randomized to Dot Diary will receive a mobile app that promotes self-management of PrEP use and sexual health. Key components include (1) a digital pill-taking and sexual diary, with pill-taking reminders; (2) sex-positive badges earned via app use; and (3) real-time feedback on protection levels afforded by PrEP. Each participant will be followed for approximately 12 months. Staff at the participating clinics will also participate in in-depth interviews to give feedback on implementation challenges and experiences in the clinic-setting, and experience working with patients using the mobile technologies.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as a cisgender man, transgender man (assigned female at birth, trans-masculine spectrum), or transgender woman (assigned male sex at birth, trans-feminine spectrum)
* Report sex with a cisgender man or transgender woman or any individual assigned male sex at birth in the past 12 months
* Age 15 years or older
* Willing and able to provide written informed consent
* Owns an iOS or Android mobile phone and able to access the internet and send and receive text messages
* Able to understand, read, and speak English or Spanish
* Newly initiated PrEP or currently on PrEP and at risk for PrEP discontinuation based on at least one of the following:

  * Initiated PrEP within the past 6 months, or
  * Has any of the following risk factors for PrEP discontinuation: missed clinic visits; age < 30; African-American or Latino; transgender gender identity; or self-reported illicit substance use

Exclusion Criteria:

* Currently enrolled in another PrEP intervention study
* Unable to complete 12 month study participation
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — cisgender man, transgender man (assigned female sex at birth, trans-masculine spectrum), or transgender woman (assigned male sex at birth, trans-feminine spectrum)
Enrollment: 300 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
PrEP adherence as measured by tenofovir diphosphate levels in dried blood spots | DBS measured through 12 months
  PrEP adherence will be measured by tenofovir diphosphate (TFV-DP) levels in dried blood spots (DBS). Adequate adherence will be defined as having a TFV-DP ≥ 700 femtomoles/punch in DBS for daily PrEP users, which has been associated with high levels of protection in prior PrEP trials.
Satisfaction with medical care | Satisfaction measured through 12 months
  Satisfaction with medical care will be measured by the Consumer Assessment of Health Care Processes and Services (CAHPS), a critical tool for evaluating patient satisfaction and patient-centeredness of care
Patient engagement | Patient engagement measured through 12 months
  Patient engagement will be measured by the short-version Patient Activation Measure (PAM).

SECONDARY OUTCOMES:
PrEP continuation based on medication refills | PrEP continuation measured through 12 months
  PrEP discontinuation will be defined as having a PrEP interruption of ≥30 days based on medication refill dates using blinded outcome ascertainment of electronic medical and pharmacy refill records.
Sexual satisfaction | Sexual satisfaction measured through 12 months
  Sexual satisfaction will be measured by the New Sexual Satisfaction Scale Short Version (NSSS-S), a validated 12-item questionnaire in which patients score their sexual satisfaction on five dimensions (sexual sensations, sexual presence/awareness, sexual exchange, emotional connection/closeness, and sexual activity)
Adherence self-efficacy | Adherence self-efficacy measured through 12 months
  Patient-reported adherence self-efficacy will be measured by the self-efficacy scale for PrEP use, which has been validated for PrEP use

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Bridge HIV, San Francisco Department of Public Health, San Francisco, California
  - San Francisco AIDS Foundation, San Francisco, California
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No